CLINICAL TRIAL: NCT00272389
Title: Prediction of Response to PEGINTERFERON and RIBAVIRIN Treatment in Patients With Chronic HCV Infection by Genetic Profile
Brief Title: Prediction of Response to Treatment of Patients With Chronic HCV Infection by Genetic Profile
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: tBEB1t-HMO-CTIL
Record Dates: First submitted 2006-01-04; First posted 2006-01-06 (Estimated); Last update posted 2006-01-06 (Estimated); Status verified 2006-01

CONDITIONS: Hepatitis C Virus Chronic Infection

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
We hypothesized that pretreatment nonresponder and responder liver tissue would show consistent differences in gene expression levels and that these differences could be used to predict treatment outcomes and this can obviate the need of the present therapeutic trial.We are interested in conducting a retrospective study using the data of patients suffering from chronic HCV infection who were treated in our department with a combination of PEGINTERFERON and RIBAVIRIN. All these patients underwent liver biopsy prior the treatment. Based on the clinical data available it is possible to determine the responders and nonresponders to this therapy.RNA will be extracted from the liver tissue and the expression of 5 genes(IFI15,IFI616,IFI1,OAS3,OAS2 )will be checked .The prediction power of the combination of these genes in differentiating responders from nonresponders will be determined.

DETAILED DESCRIPTION:
Hepatitis C virus is a leading cause of chronic liver disease, with over 170 million people infected worldwide. It is also the leading indication for liver transplantation. Complications from chronic hepatitis C infection include cirrhosis, hepatic decompensation, and hepatocellular carcinoma. As a result, treatment strategies to prevent such complications have been widely researched, although many questions remain unanswered. To date, the standard therapy for chronic hepatitis C infection is the combination of peginterferon and .ribavirin.A large proportion of patients do not respond to therapy for reasons that are unclear. The heterogeneity of viral and host phenotypes makes it unlikely that any single factor will accurately predict the cellular response to treatment.It was supposed that liver tissue of nonresponder and responder show consistent differences in gene expression levels and that these differences could be used to predict treatment outcomes.Hepatic gene expression profiling identified consistent differences in patients who subsequently fail treatment with pegylated IFN-α plus ribavirin: up-regulation of a specific set of IFN-responsive genes predicts nonresponse to exogenous therapy. These data may be of use in predicting clinical responses to treatment. 18 genes, confirmed by real-time PCR, with expression levels that differed consistently between nonresponders and responders liver tissue were detected. Levels for these 18 genes in responders liver were closer to uninfected tissue than to nonresponders liver, with a general up-regulation of gene expression in nonresponders liver. Many of these genes are IFN responsive, suggesting that the nonresponders patients have adopted a different, yet characteristic, equilibrium in their host-virus immune response(Chen L et al. Gastroentology 2005:128:1437-1444) We have found a method that can predict success or failure of the treatment of chronic hepatitis C based on the weighted expression level of a small number of genes (4-5) We derive the genes and their decision weights from the microarray data set obtained from the liver biopsy of the patients in the above mentioned paper . We would like to test the prediction power of this method in an independent set of liver tissues of treated patients in our department.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS COMPLETING TREATMENT WITH PEGINTERFERON AND RIBAVIRIN FOR CHRONIC HCV INFECTION AND UNDERWENT LIVER BIOPSY PRIOR THERAPY ONSET

Exclusion Criteria:

* TREATMENT NOT COMPLETED

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-03; Study Completion 2006-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Ilan, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Chen L, Borozan I, Feld J, Sun J, Tannis LL, Coltescu C, Heathcote J, Edwards AM, McGilvray ID. Hepatic gene expression discriminates responders and nonresponders in treatment of chronic hepatitis C viral infection. Gastroenterology. 2005 May;128(5):1437-44. doi: 10.1053/j.gastro.2005.01.059. PMID 15887125